CLINICAL TRIAL: NCT00742638
Title: An Open Label, Randomised, Valproate-Controlled Study to Evaluate the Efficiency and Safety of Quetiapine Fumarate in the Treatment of Acute Manic Patients With Bipolar Disorder.
Brief Title: To Evaluate the Efficiency and Safety of Quetiapine Fumarate in the Treatment of Acute Manic Patients With Bipolar Disorder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Yao Peifen, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00057
Record Dates: First submitted 2008-08-25; First posted 2008-08-28 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Bipolar Disorder
Keywords: CCMD-3,; CRF,; EPS,; GCP,; ICH,; ITT,; LOCF,; MADRS,; PANSS,; YMRS.; Acute; manic; patients; with; bipolar; disorder
MeSH Terms: conditions — Bipolar Disorder; Mania; Disease | interventions — Quetiapine Fumarate; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The arm 1 (Experimental): Quetiapine fumarate tablet:25mg and 200mg
  Interventions: Drug: Quetiapine fumarate
- The arm 2 (Active Comparator): Sodium valproate tablet 200mg
  Interventions: Drug: Sodium valproate

INTERVENTIONS:
Drug: Quetiapine fumarate — Investigational product: quetiapine fumarate tablet 25 mg and 200 mg
  Arms: The arm 1
Drug: Sodium valproate — Sodium valproate tablet 200 mg
  Arms: The arm 2

SUMMARY:
This is an open label, randomised, parallel-group study to compare the efficacy and safety of quetiapine and valproate used as monotherapy in the treatment of mania in patients hospitalised for an acute manic episode. After given of informed consent and undergoing screening procedures, the patients will be randomised into quetiapine or valproate group on Day 1. The efficacy of study treatment on symptoms of mania will be assessed at Day 28. Patients will not permitted to use any psychoactive or antipsychotic medications throughout the study period other than those expressly permitted by the protocol.

At each centre, the same individual will administer a specific psychiatric assessment for a patient at all study visits in order to reduce variability in rating scale scoring. Before the initiation of the study, a consistency assessment will be done among the investigators who conduct the scale assessment in each centre.

DETAILED DESCRIPTION:
The rationale for using the quetiapine to treat patients with acute mania is multifold. A potential major advantage for quetiapine is its demonstrated tolerability. Because of the low incidence of EPS, quetiapine should be better tolerated than other antipsychotic medications in this sensitive patient population. The limited potential for weight gain and prolactin elevation may promote long-term treatment compliance.

The effect of quetiapine alone or adjunctive with mood stabilizers in the treatment of acute mania in patients with bipolar disorder has been confirmed through 4 phase III clinical trials (8,9). Based on the results of these clinical trials, the use of Seroquel in the acute mania of bipolar disorder has been approved in US, UK and other major markets in Europe. Quetiapine is also been recommended as alternative therapy for acute mania treatment in the practice guideline (10). The present study is to assess the effectiveness of quetiapine and valproate in the treatment of Chinese patients with acute mania over a treatment period of 4 weeks. Primary objective The primary objective of the study is to evaluate the effectiveness of quetiapine fumarate used as monotherapy in the treatment of symptoms of acute mania in patients with bipolar disorder, by evaluation of the change from baseline in YMRS total score at Day 28 (LOCF).

Secondary objectives

The secondary objectives of the study are to evaluate the following:

* The effectiveness of quetiapine used as monotherapy to treat symptoms in patients with acute mania by evaluation of YMRS/CGI response rate at Day 28 (LOCF)
* The effectiveness of quetiapine used as monotherapy to improve clinical status in patients with acute mania by evaluation of change from baseline in CGI-S score at Day 28 (LOCF)
* The effectiveness of quetiapine used as monotherapy to treat depressive symptoms in patients with acute mania by evaluation of change from baseline in MADRS total score at Day 28 (LOCF)
* The effectiveness of quetiapine used as monotherapy to treat psychotic symptoms in patients with acute mania by evaluation of change from baseline in PANSS total score at Day 28 (LOCF)
* The safety and tolerability of quetiapine used as monotherapy to treat symptoms in patients with acute mania

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for study participation, signed by the patient's legal guardian
* Aged between 18 and 65 (inclusive)
* Is hospitalized in a psychiatric unit with an acute manic episode of bipolar disorder defined by CCMD-3 criteria i.e. [31.2] bipolar disorder whose current status is mania without psychotic symptom or [31.3] bipolar disorder whose current status is mania with psychotic symptom
* Both at screening and at randomization (Day 1), had a YMRS total score of at least 20
* Be able to understand and comply with the requirements of the study, judged by the investigator

Exclusion Criteria:

* Manic index episode judged to be the direct physiological consequence of a medical condition or treatment.
* These conditions included:

  * degenerative neurological conditions (e.g. Parkinson's disease, Huntington's disease),
  * cerebrovascular disease (e.g., stroke),
  * metabolic conditions (e.g., Vitamin B12 deficiency),
  * autoimmune conditions (e.g., systemic lupus erythematosus),
  * viral or other infections (e.g., hepatitis, mononucleosis, human immunodeficiency),
  * certain cancers.
* Manic index episode judged to be the direct physiological effect of a substance of abuse, including intoxication with or withdrawal from alcohol, amphetamine and related substances, cocaine, sedatives, hypnotics, or anxiolytics; intoxication with hallucinogens, inhalants, opioids, or phencyclidine and related substances.
* Patients who met CCMD-3 criteria for rapid cycling: at least 4 episodes of a mood disturbance in the previous 12 months that meet criteria for a hypomanic/manic or nonmajor depression/depression, or mixed episode
* Known intolerance or lack of response to quetiapine or valproate, as judged by the investigator
* Known or suspected hypersensitivity to quetiapine or valproate
* Known lack of response to clozapine
* Use of clozapine within 28 days before randomization (Day 1)
* Women in pregnancy or lactation, or female of childbearing potential without appropriate birth control measures
* Substance or alcohol dependence (except for nicotine dependence), as defined in CCMD-3, within 1 month before randomisation (Day 1).
* Continuous daily use of benzodiazepines during the month preceding screening.
* Receipt of electroconvulsive therapy (ECT) within 30 days prior to randomisation (Day 1).
* Use of antidepressant(s) during the screening period (Day -7 to Day 1) or within a period of 5 half-lives of the drug(s) prior to randomisation (Day 1).
* Use of long-acting anti-psychotic medication within 30 days prior to randomisation (Day 1)
* Thyroid-stimulating hormone concentration more than 10% above the upper limit of the normal range, regardless of treatment for hypothyroidism or hyperthyroidism.
* Use of any potent cytochrome P450 3A4 inhibitors in the 14 days preceding randomization (Day 1), e.g., ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, and saquinavir.
* Use of potent cytochrome P450 inducers (e.g. Phenytoin, carbamazepine, barbiturates, rifampin, glucocorticoids, St. John's Wort) in the 14 days preceding randomisation (Day 1).
* Renal, cardiovascular, hepatic, haematological, endocrine, congestive heart failure, or other disease or clinical finding that was unstable or in the opinion of the investigator would be negatively affected by study medication or that would affect study medication.
* Patients with diabetes mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrolment HbA1c > 8.5%
  * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks
  * Not under care of physician responsible for patient's DM care
  * Physician responsible for patient's DM care has not indicated that patient's DM is controlled
  * Physician responsible for patient's DM care has not approved patient's participation in the study
  * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 weeks
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks
* Participation in another clinical study within 4 weeks of randomisation (Day 1).
* Lack of response in previous systemic treatment with lithium and/or quetiapine.
* Medical conditions that would affect absorption, distribution, metabolism or excretion of study treatment.
* An absolute neutrophil count (ANC) of < 1.5 x 109/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-05 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The outcome measure is the change from baseline in YMRS total score at Day 28 (LOCF). | Four weeks

SECONDARY OUTCOMES:
These changes from baseline in PANSS,MADRS, CGI total score at Day 28. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China